CLINICAL TRIAL: NCT03547232
Title: Rectal Indomethacin as Early Treatment for Acute Pancreatitis (INDOMAP Trial): Study Protocol for a Multi-center, Double-blinded, Placebo-controlled, Randomized Clinical Trial
Brief Title: Rectal Indomethacin as Early Treatment for Acute Pancreatitis (INDOMAP Trial)
Acronym: INDOMAP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, DONG WU, Professor of Gastroenterology, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I-23PJ1671
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Acute Pancreatitis; Complication; Mortality Rate; Organ Failure, Multiple
Keywords: Acute pancreatitis; Indomethacin; Prognosis; Organ dysfunction
MeSH Terms: conditions — Pancreatitis; Multiple Organ Failure | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indomethacin group (Experimental): Indomethacin SR 50mg q12h from day1 to day 7 plus standard treatment for acute pancreatitis including adequate intravenous fluids, analgesics and early enteral nutrition support if possible.
  Interventions: Drug: Indomethacin SR
- Standard group (Sham Comparator): Similar shape and size suppositories without indomethacin (Placebos) given q12h from admission day 1 to day 7, plus standard treatment for acute pancreatitis including adequate intravenous fluids, analgesics and early enteral nutrition support if possible.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Indomethacin SR — Indomethacin SR 50mg given q12h from admission day 1 to day 7
  Other Names: YINDUOMEIXIN
  Arms: Indomethacin group
Drug: Placebos — Similar shape and size suppositories (Placebos) without indomethacin given q12h from admission day 1 to day 7
  Other Names: SHAM
  Arms: Standard group

SUMMARY:
Acute pancreatitis (AP) is an inflammatory condition of the pancreas following the activated pancreatic enzymes induced by varied causes, with or without other organ(s) dysfunction. The production and release of inflammatory factors is generally considered as the key factor of pathogenesis. Non-steroidal anti-inflammatory drugs (NSAIDs) are the most commonly applied agents for inflammatory diseases. A series studies have proved that indomethacin can reduce the risk of post-endoscopic retrograde cholangiopancreatography (ERCP), but high-quality evidence is still lacking in the field of effectiveness of NSAIDs to treat, rather than prevent, other types of AP. Majority of animal experiments showed that NSAIDs had protective effects for organ functions, but the results of several preliminary clinical studies were inconsistent. Randomized controlled trials are eagerly awaited to elucidate its effects on AP.

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 18-80 years with a diagnosis of AP based on at least 2 of the following criteria:
* Abdominal pain characteristic of AP
* Serum amylase and/or lipase ≥ 3 times the upper limit of normal
* Characteristic findings of AP on abdominal CT scan will be screened for study enrollment.

Exclusion Criteria:

* Onset time >24 hours
* Presence of renal dysfunction (serum creatinine > 1.5 *normal upper limit)
* Severe liver dysfunction
* Active peptic ulcer disease or GI bleeding
* Pregnancy or breast-feeding
* Hypersensitivity to NSAIDs
* New-onset, exacerbation or uncontrolled hypertension
* Presence of serious cardiovascular events, including severe heart failure, myocardial infarction (MI) and stroke
* Mental disability
* Malignancy-associated acute pancreatitis
* Post-ERCP pancreatitis
* Informed consent not signed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1504 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurence rate of organ dysfunction caused by acute pancreatitis | 1 week
  Accumulation of varied organ dysfunction, especially the cardiovascular, renal and respiratory systems

SECONDARY OUTCOMES:
Occurence rate of pancreatic necrosis | 1 month
  Accumulation of the key local complication of acute pancreatitis
Incidence rate of ICU admission | 1 month
  Evaluation of critical severe acute pancreatitis
Mortality | 1 month
  The number of deaths during a particular period of time

OTHER OUTCOMES:
Hospitalization cost | 1 month
  Expense of acute pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wu, M.D., Study Chair — Peking Union Medical College Hospital; Zhitao Lu, M.D., Principal Investigator — Baoding Seventh Hospital; Yanfeng Wang, M.D., Principal Investigator — Liangxiang Hospital; Shanshan Yu, M.D., Principal Investigator — Guiyang Second People's Hospital; Na Wu, M.D., Principal Investigator — Dengzhou People's Hospital; Mei Liu, M.D., Principal Investigator — Affiliated Hospital of Qinghai University; Xiao Fan, M.D., Principal Investigator — Second People Hospital of Nanyang; Zuoyan Wu, MD, Principal Investigator — Peking University Sixth Hospital; Ruifeng Wang, MD, Principal Investigator — Harbin Medical University; Baofeng Zhu, MD, Principal Investigator — Nantong First People's Hospital; Yan Shi, MD, Principal Investigator — The Second People's Hospital of Huai'an; Ming Sun, MD, Principal Investigator — Suqian People's Hospital; Wei Huang, MD, Principal Investigator — Wuxi Third People's Hospital; Shicheng Zheng, MD, Principal Investigator — West China Longquan Hospital Sichuan University; Jianzhong Yang, MD, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Daoyuan Jing, MD, Principal Investigator — Jinhua Municipal Central Hospital; Hong Liu, MD, Principal Investigator — Lishui Municipal Central Hospital
Locations (17):
- China (17):
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Liangxiang Hospital, Beijing, Beijing Municipality
  - Guiyang Second People's Hospital, Guiyang, Guizhou
  - Baoding Seventh Hospital, Baoding, Hebei
  - Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Dengzhou People's Hospital, Dengzhou, Henan
  - Second People Hospital of Nanyang, Nanyang, Henan
  - The Second People's Hospital of Huai'an, Huaian, Jiangsu
  - Nantong First People's Hospital, Nantong, Jiangsu
  - Suqian People's Hospital, Suqian, Jiangsu
  - Wuxi Third People's Hospital, Wuxi, Jiangsu
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - West China Longquan Hospital Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Lishui Municipal Central Hospital, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorsky VA, Agapov MA, Khoreva MV, Leonenko IV. The effect of lornoxicam on TLR2 and TLR4 messenger RNA expression and tumor necrosis factor-alpha, interleukin-6, and interleukin-8 secretion in patients with systemic complications of acute pancreatitis. Pancreas. 2015 Jul;44(5):824-30. doi: 10.1097/MPA.0000000000000344. PMID 25872171
- See also: A small sample study of NSAIDs for treatment of acute pancreatitis — https://www.ncbi.nlm.nih.gov/pubmed/?term=25872171